CLINICAL TRIAL: NCT03848728
Title: Strategic Antiretroviral Therapy and HIV Testing for Youth in Rural Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Infectious Diseases Research Collaboration, Uganda (Other); Kenya Medical Research Institute (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SEARCH Youth; UG3HD096915 (NIH); UH3HD096915 (NIH)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: HIV
Keywords: HIV; Adolescent; Young Adult; Viral Load; Counseling; Costs and Cost Analysis

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Clinics (Experimental): SEARCH Youth combination intervention, which includes life-stage assessment and counseling, rapid VL feedback, structured choice clinic access, and e-collaboratives chat-based discussion among providers
  Interventions: Other: SEARCH Youth combination intervention
- Control Clinics (No Intervention): Optimized country standard of care

INTERVENTIONS:
Other: SEARCH Youth combination intervention — * Administration of life-stage assessment tool
  * Structured choice clinic access
  * Rapid feedback of VL results
  * Provider e-collaboratives with chat groups for discussions of challenging cases using de-identified information
  Arms: Intervention Clinics

SUMMARY:
The goal of this study is to evaluate the effect of a combination intervention on long-term HIV viral load (VL) suppression among HIV-infected adolescents and young adults 15-24 years of age. The study will take place in 28 rural HIV clinics in western Kenya and southwest Uganda. Clinics will be randomly chosen to either continue to provide study participants standard care or to provide the study intervention, which consists of discussion and counseling on major issues or life events, flexible access to the clinic, and rapid turnaround of VL test results. Participants will take part in the study for at least 2 years.

DETAILED DESCRIPTION:
The randomized controlled trial (RCT) will evaluate the effect of the SEARCH Youth intervention on long-term HIV viral load suppression among HIV-infected adolescents/young adults. The study's intervention is based on the PRECEDE model of behavioral change that is targeted towards adolescent and young adult behavior. The study design is a cluster-randomized trial where the unit of randomization is the HIV clinic: 14 clinics randomized to the intervention and 14 to the optimized country standard of care (Differentiated ART care, standard clinic hours, routine VL monitoring, access to 2nd and 3rd line ART), balanced within country. The target enrollment for the intervention is approximately 2300 (50-100 adolescents/young adults with HIV in each clinic, plus family members, providers and others taking part in qualitative interviews).

Community-tailored youth testing and linkage strategies for ART will be implemented to recruit youth for the SEARCH Youth combination intervention RCT. Strategies to reach youth at the highest risk of HIV infection will be implemented. Those individuals who test HIV-positive will be referred to the local clinic for HIV treatment services and, if they otherwise meet entry criteria, to the SEARCH Youth study for possible inclusion.

The components of the SEARCH Youth intervention include:

* Administration of life-stage assessment tool at the beginning of each visit that links to life-stage specific actions and puts subsequent medical discussions into an appropriate context
* Structured choice clinic access which will provide a choice to schedule visits during or after routine clinic hours or in an alternate location, with some phone-only visits available between in-person visits
* Rapid feedback of VL results, by phone or in person, aiming to be provided within 72 hours, to provide immediate feedback on HIV suppression and engage participants in their overall health
* Provider e-collaboratives that comprises of chat groups using WhatsApp or similar secure messaging applications to solicit input about challenging cases using de-identified information

Participants will take part in the study for at least 2 years.

Some participants, family members, providers, HIV-negative youth and key informants will also take part in qualitative interview guides. Costs of the SEARCH Youth intervention will be evaluated to assess its efficiency and cost-effectiveness including as cost per participant, cost per additional participant with viral suppression and cost per DALY gained.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection diagnosed according to country testing guidelines
* Age 15-24 years
* Enrolled in care in a study clinic
* Ability and willingness to provide informed consent

Exclusion Criteria:

* None

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1988 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane V Havlir, MD, Principal Investigator — University of California, San Francisco; Moses R Kamya, MBChB, MMed, PhD, Principal Investigator — Makerere University
Locations (2):
- Western Kenya, Sindo, Kenya
- Southwestern Uganda, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamb MR, Fayorsey R, Nuwagaba-Biribonwoha H, Viola V, Mutabazi V, Alwar T, Casalini C, Elul B. High attrition before and after ART initiation among youth (15-24 years of age) enrolled in HIV care. AIDS. 2014 Feb 20;28(4):559-68. doi: 10.1097/QAD.0000000000000054. PMID 24076661
- [Background] Evans D, Menezes C, Mahomed K, Macdonald P, Untiedt S, Levin L, Jaffray I, Bhana N, Firnhaber C, Maskew M. Treatment outcomes of HIV-infected adolescents attending public-sector HIV clinics across Gauteng and Mpumalanga, South Africa. AIDS Res Hum Retroviruses. 2013 Jun;29(6):892-900. doi: 10.1089/AID.2012.0215. Epub 2013 Feb 25. PMID 23373540
- [Background] Nachega JB, Hislop M, Nguyen H, Dowdy DW, Chaisson RE, Regensberg L, Cotton M, Maartens G. Antiretroviral therapy adherence, virologic and immunologic outcomes in adolescents compared with adults in southern Africa. J Acquir Immune Defic Syndr. 2009 May 1;51(1):65-71. doi: 10.1097/QAI.0b013e318199072e. PMID 19282780
- [Background] Jobanputra K, Parker LA, Azih C, Okello V, Maphalala G, Kershberger B, Khogali M, Lujan J, Antierens A, Teck R, Ellman T, Kosgei R, Reid T. Factors associated with virological failure and suppression after enhanced adherence counselling, in children, adolescents and adults on antiretroviral therapy for HIV in Swaziland. PLoS One. 2015 Feb 19;10(2):e0116144. doi: 10.1371/journal.pone.0116144. eCollection 2015. PMID 25695494
- [Background] Zurcher K, Mooser A, Anderegg N, Tymejczyk O, Couvillon MJ, Nash D, Egger M; IeDEA and MESH consortia. Outcomes of HIV-positive patients lost to follow-up in African treatment programmes. Trop Med Int Health. 2017 Apr;22(4):375-387. doi: 10.1111/tmi.12843. Epub 2017 Feb 20. PMID 28102610
- [Background] Massaquoi M, Zachariah R, Manzi M, Pasulani O, Misindi D, Mwagomba B, Bauernfeind A, Harries AD. Patient retention and attrition on antiretroviral treatment at district level in rural Malawi. Trans R Soc Trop Med Hyg. 2009 Jun;103(6):594-600. doi: 10.1016/j.trstmh.2009.02.012. Epub 2009 Mar 18. PMID 19298993
- [Derived] Ruel T, Mwangwa F, Balzer LB, Ayieko J, Nyabuti M, Mugoma WE, Kabami J, Kamugisha B, Black D, Nzarubara B, Opel F, Schrom J, Agengo G, Nakigudde J, Atuhaire HN, Schwab J, Peng J, Camlin C, Shade SB, Bukusi E, Kapogiannis BG, Charlebois E, Kamya MR, Havlir D. A multilevel health system intervention for virological suppression in adolescents and young adults living with HIV in rural Kenya and Uganda (SEARCH-Youth): a cluster randomised trial. Lancet HIV. 2023 Aug;10(8):e518-e527. doi: 10.1016/S2352-3018(23)00118-2. PMID 37541706
- [Derived] Johnson-Peretz J, Lebu S, Akatukwasa C, Getahun M, Ruel T, Lee J, Ayieko J, Mwangwa F, Owino L, Onyango A, Maeri I, Atwine F, Charlebois ED, Bukusi EA, Kamya MR, Havlir DV, Camlin CS. "I was still very young": agency, stigma and HIV care strategies at school, baseline results of a qualitative study among youth in rural Kenya and Uganda. J Int AIDS Soc. 2022 Jul;25 Suppl 1(Suppl 1):e25919. doi: 10.1002/jia2.25919. PMID 35818888
- [Derived] Mwangwa F, Charlebois ED, Ayieko J, Olio W, Black D, Peng J, Kwarisiima D, Kabami J, Balzer LB, Petersen ML, Kapogiannis B, Kamya MR, Havlir DV, Ruel TD. Two or more significant life-events in 6-months are associated with lower rates of HIV treatment and virologic suppression among youth with HIV in Uganda and Kenya. AIDS Care. 2023 Jan;35(1):95-105. doi: 10.1080/09540121.2022.2052260. Epub 2022 May 16. PMID 35578398

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics
Groups:
- Intervention Clinics: SEARCH Youth combination intervention, which includes life-stage assessment and counseling, rapid VL feedback, structured choice clinic access, and e-collaboratives chat-based discussion among providers
  SEARCH Youth combination intervention:
  * Administration of life-stage assessment tool
  * Structured choice clinic access
  * Rapid feedback of VL results
  * Provider e-collaboratives with chat groups for discussions of challenging cases using de-identified information
Period: Overall Study
Arm/Group | Intervention Clinics | Control Clinics
Started | 1012; 14 Clinics | 976; 14 Clinics
Completed | 865; 14 Clinics | 809; 14 Clinics
Not Completed | 147; 0 Clinics | 167; 0 Clinics
Not completed — Death | 16 | 13
Not completed — Outmigrated to non-study community | 98 | 106
Not completed — Transfered to non-study clinic | 32 | 48
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population includes participants who were included in the primary analysis, enrolled before December 1, 2019.
Groups:
- Intervention Clinics: SEARCH Youth combination intervention, which includes life-stage assessment and counseling, rapid VL feedback, structured choice clinic access, and e-collaboratives chat-based discussion among providers
  SEARCH Youth combination intervention:
  * Administration of life-stage assessment tool
  * Structured choice clinic access
  * Rapid feedback of VL results
  * Provider e-collaboratives with chat groups for discussions of challenging cases using de-identified information
  Information presented for participants included in primary analysis.
- Control Clinics: Optimized country standard of care.
  Information presented for participants included in primary analysis.
- Total: Total of all reporting groups
Arm/Group | Intervention Clinics | Control Clinics | Total
Number analyzed (Participants) | 785 | 764 | 1549
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Median age | 21 [19 to 23] | 21 [19 to 23] | 21 [19 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 643 | 605 | 1248
  Male | 142 | 159 | 301
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/Black | 785 | 764 | 1549
Region of Enrollment [Number; unit: participants]
  Uganda | 332 | 324 | 656
  Kenya | 453 | 440 | 893
Education (started or completed) [Count of Participants; unit: Participants]
  No school | 31 | 24 | 55
  Primary school | 507 | 525 | 1032
  Secondary school | 194 | 175 | 369
  Tertiary school | 53 | 40 | 93
  At boarding school | 56 | 56 | 112
Employment status [Count of Participants; unit: Participants]
  Employed | 283 | 308 | 591
  In school | 165 | 155 | 320
  Unemployed | 337 | 301 | 638
Marital status [Count of Participants; unit: Participants]
  Single, never married | 342 | 291 | 633
  Married, monogamous | 306 | 327 | 633
  Married, polygamous | 44 | 51 | 95
  Widowed | 3 | 6 | 9
  Divorced | 90 | 89 | 179
Number of children [Count of Participants; unit: Participants]
  0 children | 330 | 323 | 653
  1 child | 258 | 227 | 485
  2 children | 129 | 131 | 260
  3-5 children | 51 | 64 | 115
Drinks alcohol [Count of Participants; unit: Participants] | 137 | 94 | 231
Mobile [Count of Participants; unit: Participants] — Lived away from home for more than 1 month in the previous 6 months.
  Participants | 210 | 229 | 439
Antiretroviral regimen at enrolment [Count of Participants; unit: Participants] — Population: Data missing from 16 participants - 7 in intervention group, 9 in control group
  Participants
    number analyzed (Participants) | 778 | 755 | 1533
    TDF-3TC-EFV | 591 | 527 | 1118
    TDF-3TC-DTG | 81 | 101 | 182
    AZT-3TC-NVP | 33 | 42 | 75
    TDF-3TC-ATV/r | 10 | 18 | 28
    AZT-3TC-ATV/r | 12 | 14 | 26
    ABC-3TC-EFV | 12 | 11 | 23
    Other | 39 | 42 | 81
Baseline viral load <400 copies per mL [Count of Participants; unit: Participants] — Population: Data missing from 16 participants: 5 intervention participants, 11 control participants
  Participants
    number analyzed (Participants) | 780 | 753 | 1533
    (all) | 573 | 574 | 1147
Baseline care status [Count of Participants; unit: Participants] — Population: Data missing for 2 participants, 1 intervention participant, 1 control participant
  Participants
    number analyzed (Participants) | 784 | 763 | 1547
    Recently engaged - started treatment within 6 months of enrolment | 252 | 214 | 466
    Engaged - started treatment > 6 months before enrolment with HIV care visit within 6 months | 496 | 530 | 1026
    Re-engaging - started treatment > than 6 months before enrolment, no HIV care visit within 6 months | 36 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of SEARCH Youth Intervention
Description: Percentage of study participants with virologic suppression (HIV RNA <400 c/mL) at 2 years of follow-up. Mean was calculated as the average percentage across the clusters (clinics)
Time Frame: 2 years
Population: Study participants at year 2, excluding those who enrolled on/after Dec 1, 2019, transferred care, outmigrated, or withdrew.
Measure: Mean (95% Confidence Interval); unit: % of participants
Units Other Than Participants: Clinics
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | 785 | 764
Number analyzed (Clinics) | 14 | 14
% of participants
  All | 88.2 [84.8 to 91.7] | 80.5 [76.9 to 84.1]
  Engaged: number analyzed (Participants) | 496 | 530
  Engaged | 90.9 [87.7 to 94.0] | 85.3 [81.0 to 89.5]
  Recently engaged: number analyzed (Participants) | 252 | 214
  Recently engaged | 80.1 [72.7 to 87.5] | 73.5 [67.1 to 79.8]
  Re-engaging: number analyzed (Participants) | 36 | 19
  Re-engaging | 84.8 [72.7 to 97.0] | 53.2 [29.5 to 76.9]
Statistical Analysis 1: Comparison: Intervention Clinics vs Control Clinics; Test type: Superiority; p = 0.0019, TMLE; Risk Ratio (RR) = 1.10, 95% CI 2-sided [1.03 to 1.16]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Non-fatal serious adverse events were reported regardless of relationship to the study intervention in the intervention arm only. Control arm participants were not contacted during the study except at baseline and endpoint. Other [Not Including Serious] Adverse Events were not monitored/assessed in both intervention and control arms. Fatal serious adverse events were reported in both the intervention arm and the control arm regardless of relationship.
Arm/Group | Intervention Clinics | Control Clinics
All-Cause Mortality (participants affected / at risk) | 16/1012 | 13/976
Serious Adverse Events (participants affected / at risk) | 48/1012 | 13/976
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Intervention Clinics (N=1012) | Control Clinics (N=976)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Urinary tract infection (Infections and infestations) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Hernia (Gastrointestinal disorders) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Malaria (Infections and infestations) | 4 (4) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Depression (Psychiatric disorders) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Pneumonia (Infections and infestations) | 2 (2) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Oral thrush (Infections and infestations) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Cesarean infant delivery (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Anemia (Blood and lymphatic system disorders) | 5 (6) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Typhoid fever (Infections and infestations) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Seizures (Nervous system disorders) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Suspected bacterial or tubercular respiratory infection resulting in death (Infections and infestations) | 1 (1) | 0 (0)
Liver disease resulting in death (Hepatobiliary disorders) | 1 (1) | 0 (0)
Presumed sepsis resulting in death (Immune system disorders) | 1 (1) | 0 (0)
Respiratory failure resulting in death (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hepatocellular carcinoma resulting in death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death, cause unknown (General disorders) | 3 (3) | 1 (1)
Suspected tuberculosis resulting in death (Infections and infestations) | 1 (1) | 0 (0)
Severe anemia resulting in death (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
AIDS resulting in death (Immune system disorders) | 0 (0) | 2 (2)
Kidney disease resulting in death (Renal and urinary disorders) | 0 (0) | 1 (1)
Sickle cell anemia resulting in death (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Severe malnutrition resulting in death (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary tuberculosis resulting in death (Infections and infestations) | 1 (1) | 2 (2)
Organ failure, cause unknown, resulting in death (General disorders) | 0 (0) | 1 (1)
Threatened abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
Encephalitis (Infections and infestations) | 1 (1) | 0/0 (0) — Serious Adverse Events not resulting in death were not monitored/assessed in the control arm.
CNS-TB with possible brain tumor resulting in death (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure resulting in death (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal tumor resulting in death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pre-eclampsia toxemia resulting in death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Kaposi sarcoma resulting in death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia resulting in death (Infections and infestations) | 0 (0) | 1 (1)
Complications following Cesarean childbirth resulting in death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03848728/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT03848728/SAP_001.pdf
  • Informed Consent Form (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT03848728/ICF_002.pdf